



## **STATISTIC ANALYSIS**

## Title

Influence of residual astigmatism on visual acuity in patients undergoing cataract surgery with trifocal intraocular lens implantation

Approved by the CEIm Grupo Hospitalario Quirónsalud-Catalunya on July 29, 2019 (ID: 2019/65-OFT-CMT)



## **Analysis of results**

The data will be exported to a database expressly built for this project with the security guarantees that guarantee compliance with the data protection laws in force. Information will be obtained from a minimum of 48 patients. The IBM® SPSS® Statistics v26 statistical program will be used to perform descriptive analysis and inferential analysis. The Kolmogorov-Smirnov / Shapiro-Wilk test, graphical tests based on the Q-Q Plot, and Normal-Plot normality graphs will be used as sample normality tests. Quantitative variables will be expressed as mean and standard deviation. For the inference of parameters, the hypothesis contrast tests and appropriate confidence intervals will be used in each case: t-Student, ANOVA, and their non-parametric equivalents when necessary (Wilcoxon signed-rank test, Kruskal-Wallis test). The level of significance in all analyzes will be p <0.05.